CLINICAL TRIAL: NCT05606263
Title: Efficacy and Safety of Caldonirimab Plus Nimotuzumab for Recurrent or Metastatic Cervical Cancer: a Multicenter, Single-arm, Prospective Phase II Trial
Brief Title: Efficacy and Safety of Caldonirimab Plus Nimotuzumab for Recurrent or Metastatic Cervical Cancer
Acronym: GCR-05
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Liu Zi, Professor, Xi'an Jiaotong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCR-5
Record Dates: First submitted 2022-10-31; First posted 2022-11-04 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; Caldonirimab; Nimotuzumab
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — nimotuzumab

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Caldonirimab and nimotuzumab (Experimental): Caldonirimab combined with nimotuzumab therapy
  Interventions: Drug: Caldonirimab and Nimotuzumab

INTERVENTIONS:
Drug: Caldonirimab and Nimotuzumab — Subjects will receive caldonirimab (6mg/Kg, q2w) until disease progression or for a maximum of 12 months, and Nimotuzumab (400mg/time, q2w) for a total of 8 cycles

SUMMARY:
To evaluated the efficacy and safety of caldonirimab plus nimotuzumab as second-line or later therapy for recurrent or metastatic cervical cancer

DETAILED DESCRIPTION:
Caldonirimab, a PD-1/CTLA-4 bispecific antibody, has shown promising efficacy and tolerable toxicity in the first-line treatment of recurrent or metastatic cervical cancer. In this study, patients with recurrent or metastatic cervical cancer, after failure of first-line platinum-containing chemotherapy or intolerance to chemotherapy, will be included in this study according to the prescribed criteria in the protocal. Nimotuzumab 400 mg/time, intravenous injection, q2w, a total of 8 times; Caldonirimab 6 mg/Kg, q2w. Assess objective response rate; disease control rate; duration of overall response and safety ( adverse event).

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 & ≤80.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 2.
3. Subjects must have histologically or cytologically confirmed recurrent or metastatic carcinoma of the cervix
4. Patients have received at least one systemic therapy or who cannot tolerate chemotherapy in the recurrent or metastatic setting
5. Has at least one measurable lesion based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 assessed by investigator.
6. Has adequate organ function.
7. Life expectancy ≥3 months.

Exclusion Criteria:

1. Concurrent enrollment in another clinical study;
2. Clinically significant hydronephrosis, as determined by the investigator, not alleviated by nephrostomy or ureteral stent;
3. Had received caldonirimab or nimotuzumab before;
4. Known history of testing positive for human immunodeficiency virus (HIV) or known active acquired immunodeficiency syndrome.
5. Known active hepatitis B or C infections (known positive hepatitis B surface antigen [HBsAg] result or positive hepatitis C virus [HCV] antibody with detectable HCV ribonucleic acid [RNA] results).
6. Patients with clinically significant cardio-cerebrovascular disease
7. Known allergy or reaction to any component of the two drugs.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 2 years
  ORR is defined as the proportion of subjects with confirmed CR or PR, based on RECIST v1.1

SECONDARY OUTCOMES:
Disease control rate (DCR) | 2 years
  The DCR is defined as the proportion of subjects with CR, PR, or SD, based on RECIST 1.1
Duration of response (DoR) | 2 years
  Duration of response is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first
Progression-free survival (PFS) | 2 years
  Progression-free survival is defined as the time from the start of treatment with caldonirimab and nimotuzumab until the first documentation of disease progression or death due to any cause, whichever occurs first
Adverse events (AEs) | 90 days
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Zi Liu, Principal Investigator — Xi'an Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xi'an Jiao Tong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No